CLINICAL TRIAL: NCT03511794
Title: Effectiveness of the Hepatitis B Vaccine Post-Hematopoietic Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918085; 18-H-N085
Record Dates: First submitted 2018-04-27; First posted 2018-04-30 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Hepatitis B
Keywords: Hepatitis B Reactivation; Allogenic Stem Cell Transplant; Natural History
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hep B vaccine: 1. Patient must have received at least one dose of the hepatitis B vaccine

SUMMARY:
Background:

Stem cell transplants (SCTs) are important in treating many diseases. There are two main types of transplants. Autologous stem cells come from the person getting the cells. Allogeneic stem cells come from another person. The risk of hepatitis B virus (HBV) is high after allogeneic SCT. Even if a person receives the HBV vaccine after transplant, he or she may not really be immune to HBV. The person may become immune only after repeated series of the vaccine. Researchers need to learn more about the HBV vaccine in people after transplant so it can be most effective.

Objective:

To assess the rate of achieved HBV immunity for people who had an SCT who did not become immune with the first vaccine series and require 2 or more series.

Eligibility:

People who have had at least 1 dose of the HBV vaccine and were enrolled in these protocols: 99-H-0050, 10-H-0154, and 08-H-0046

Design:

Participants will be screened in the other protocols.

Participants data and medical charts will be reviewed.

Data from up to 350 participants who had transplants before March 2016 will be reviewed.

Participants data will be collected:

Demographic data

Type of transplant

Type of donor

Clinical information about the transplant...

DETAILED DESCRIPTION:
Based on current medical literature, the risk of hepatitis B reactivation is high after allogenic stem cell transplant and can be a major problem in the post-transplant population, leading to increased morbidity and mortality. Additionally, many people in the general population and transplant population do not achieve immunity against hepatitis B with the first vaccination series and may require repeat series.

Currently, it is unclear as to what percentage of post-transplant patients have a failed or delayed immunity against hepatitis B and how many vaccine series it may take to eventually achieve immunity. Previous data has eluded toward a seroconversion rate of 64% in children and adults after vaccination with 20% of patients losing immunity by 5-years post-vaccination. Additionally, the study found that 25% of patients did not achieve protective titers following one vaccination series and of those that went on to be revaccinated, 55% achieved seroconversion.

This is a single-center, retrospective analysis examining the effectiveness of the hepatitis B vaccine posthematopoietic stem cell transplant and the impact of factors that may affect seroconversion. Through this study, we hope to collect data on hepatitis B vaccination and recommend potential protocol revisions if trends are found. We hypothesize that hepatitis B immunity post-first vaccine series will occur in the majority of patients evaluated and that patients failing to respond to the first vaccine series, will respond to subsequent vaccination series.

The primary objective will be to assess the rate of achieved immunity for those patients that do not achieve immunity with the first vaccine series and require two or more vaccine series. Secondary and exploratory objectives will include the evaluation of the percentages of patients responding to vaccination on the 1st, 2nd, and 3rd attempt at the hepatitis B vaccination series, the rate of reactivation of hepatitis B, and the analysis of factors potentially impacting the response to vaccination.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patient must have received at least one dose of the hepatitis B vaccine and been enrolled in the following NHLBI protocols: 99-H-0050, 10-H-0154, and 08-H-0046.
  2. Post-vaccination titers must be available for patients included in the study.

EXCLUSION CRITERIA:

1. No post-vaccination titers available.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who have received at least one dose of the hepatitis B vaccine
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
to assess the rate of achieved immunity for those patients that do not achieve immunity with the first vaccine series and require two or more vaccine series | 6 months
  to assess the rate of achieved immunity for those patients that do not achieve immunity with the first vaccine series and require two or more vaccine series

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States